CLINICAL TRIAL: NCT02565355
Title: Randomized Controlled Trial of Food Elimination Based on IgG Antibodies for Treatment of Functional Gastrointestinal Diseases (FGIDs) in Children
Brief Title: Targeted Food Elimination for Treatment of Functional Gastrointestinal Diseases in Children
Acronym: FGID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: University of Western Ontario, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 106580
Record Dates: First submitted 2015-09-09; First posted 2015-10-01 (Estimated); Last update posted 2017-10-03 (Actual); Status verified 2017-08

CONDITIONS: Functional Gastrointestinal Disorders; Functional Abdominal Pain Syndrome; Abdominal Pain (AP)
Keywords: Pediatric Gastroenterology
MeSH Terms: conditions — Gastrointestinal Diseases; Abdominal Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Modification/Dietary Exclusion (Other): In the lifestyle modification group, where specific IgG antibodies to foods are identified, the intervention is appropriate dietary elimination. The IgG antibody results will be disclosed and specific dietary elimination advice will be provided by an experienced dietician; provide diet alternatives to prevent nutritional deficiencies and improve adherence to diet. To improve compliance, a maximum of 2 high IgG positive foods will be eliminated at any one time in each 4 week period. Children will be followed-up in PG clinic at 4-weekly intervals for 16 weeks. Response is defined as more than 50% improvement in frequency and severity of abdominal pain. They will be assessed at visits 2, 3, 4 and 5 for follow-up, and non-responders, will cross over to the other arm of the study.
  Interventions: Other: Dietary Exclusion
- The Standard Treatment Group (Other): The standard therapy group will not receive results of IgG antibody testing. The patients will receive conventional treatment for Abdominal Pain as per usual practice at the Pediatric GI (PG) Clinic - counseling, reassurance, improving coping strategies and pain relief as appropriate. Children will be followed-up in PG clinic at 4-weekly intervals for 16 weeks. Response is defined as more than 50% improvement in frequency and severity of abdominal pain. They will be assessed at visits 2, 3, 4 and 5 for follow-up, and non-responders, will cross over to the other arm of the study.
  Interventions: Other: Standard Treatment

INTERVENTIONS:
Other: Dietary Exclusion — The IgG antibody results will be disclosed ONLY to the patients in the lifestyle modification group by phone approximately one week after clinic visit.. 'Dietary Exclusion' will be advised by a dietitian. Patients are advised to eliminate a maximum of two foods as identified by high IgG antibody titres.
  Arms: Lifestyle Modification/Dietary Exclusion
Other: Standard Treatment — The standard therapy group will receive conventional treatment for Abdominal Pain as per usual practice at the Pediatric GI (PG) Clinic - counseling, reassurance, improving coping strategies and pain relievers as appropriate.
  Arms: The Standard Treatment Group

SUMMARY:
Recurrent Abdominal Pain (RAP) in children is common and causes significant functional impairment and poor quality of life. Lifestyle factors such as diet, anxiety, and stress are important triggers of abdominal pains, but there is lack of high quality research evidence on optimal treatment modalities in children. This study aims to evaluate the effect of food elimination on abdominal pain frequency and severity in a cohort of children with abdominal pain associated Functional Gastrointestinal Diseases (FGID). The primary outcome will be a comparison of abdominal pain frequency and severity between standard therapy and targeted food elimination, based on IgG antibody results to a multiple food antigen panel. The investigators anticipate that 'targeted dietary elimination' as a treatment strategy will resolve abdominal pain and improve quality of life in children.

DETAILED DESCRIPTION:
Randomized controlled single center trial. Setting: Outpatient pediatric gastroenterology (PG) clinic, Children's Hospital, London, Canada. Methodology: After a 4 week run in period, 60 children aged 5-18 years, meeting Rome 3 inclusion criteria for abdominal pain associated FGID will be recruited to the trial. After informed consent, the participants will be randomized to either a standard treatment or lifestyle modification (dietary elimination) group in the ratio of 1:1. IgG testing to food antigens will be completed in both groups using a commercially available specific IgG ELISA-based multiple food allergen panel but will ONLY be disclosed for the lifestyle modification group. The patient will receive specific advice by a dietitian to exclude a maximum of two food items from his/her diet for 4 weeks. Children will be followed-up in PG clinic at 4-weekly intervals for 16 weeks. At every clinic visit, Diary of food intake, Abdominal Pain Index (API) and Quality of Life (QOL) questionnaire will be completed by both child and parent. The standard therapy group will receive conventional treatment for Abdominal Pain (AP) as per usual practice at the PG Clinic. Response is defined as more than 50% improvement in frequency and severity of abdominal pain. At each follow up visit, non-responders will cross over to the other arm of the study. At the end of the trial, non-responders in either group will continue to receive conventional treatment in the PG Clinic. Responders will be discharged back to their family physicians. Data will be analyzed using IBM SPSS Statistics, version 22.0.

ELIGIBILITY:
Inclusion Criteria:

1. Children 5-18 years of age with a diagnosis of Abdominal Pain-related FGIDs (Functional Abdominal Pain , FAP syndrome, Functional Dyspepsia, Irritable Bowel Syndrome, Abdominal Migraine) as defined by the Rome 3 criteria.
2. Acquisition of informed consent

Exclusion Criteria:

1. Children less than 5 years of age
2. Organic cause of abdominal pain established by investigations (e.g. Crohn's disease)
3. Diagnosis of failure-to-thrive or co-morbid chronic physical disease (e.g., Diabetes)
4. Any medical condition that in the opinion of the investigator would be unsafe for trial participation.
5. Lack of follow-up or failure to comply with study procedures.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Abdominal Pain Index: Child Form and Parent Proxy Form | 4 week run in period to Visit 5 (Week 16)
  Primary Outcome: The Abdominal Pain (AP) frequency and severity is calculated in each clinic visit using a 4 point questionnaire - the validated Abdominal Pain Index (API): Child Form and Parent Proxy form for age range 8 to 18 years. For age range 5 to 7 years, only the Abdominal Pain Index: Parent proxy form will be used. The 4 point scale measures the frequency of abdominal pain (Scores range 0-none to 5-every day and constant), duration of abdominal pain (scores range 0-no pain to 5-all day) and severity of abdominal pain (scores range from 0-no pain to 10-most pain). Improvement in AP is defined as >50% reduction in frequency and severity of AP in food elimination and standard treatment groups.

SECONDARY OUTCOMES:
KINDL Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents | 4 week run in period to Visit 5 (Week 16)
  The KINDL Questionnaire: self report and parent proxy versions will be used for different age groups. The KINDL questionnaire consists of 24 Likert-scaled items associated with six dimensions:physical well-being, emotional well-being, self-esteem, family, friends and everyday functioning (school or nursery school/kindergarten). The sub-scales of these six dimensions can be combined to produce a total score.
Patient Compliance | 4 week run in period to Visit 5 (Week 16)
  Compliance with dietary exclusion in dietary exclusion group at visits 3, 4 and 5. Compliance with conventional treatment in standard group at visits 3, 4 and 5. Adherence to advice and treatment will be measured by clinician impression at visits in both groups. (measured by consistency of completion of diaries and patient reporting of adherence to medical advice).

CONTACTS AND LOCATIONS:
Overall Officials: Dhandapani Ashok, MD, Principal Investigator — Children's Hospital of Western Ontario

REFERENCES:
- [Background] Rasquin A, Di Lorenzo C, Forbes D, Guiraldes E, Hyams JS, Staiano A, Walker LS. Childhood functional gastrointestinal disorders: child/adolescent. Gastroenterology. 2006 Apr;130(5):1527-37. doi: 10.1053/j.gastro.2005.08.063. PMID 16678566
- [Background] Miele E, Simeone D, Marino A, Greco L, Auricchio R, Novek SJ, Staiano A. Functional gastrointestinal disorders in children: an Italian prospective survey. Pediatrics. 2004 Jul;114(1):73-8. doi: 10.1542/peds.114.1.73. PMID 15231910
- [Background] Crandall WV, Halterman TE, Mackner LM. Anxiety and pain symptoms in children with inflammatory bowel disease and functional gastrointestinal disorders undergoing colonoscopy. J Pediatr Gastroenterol Nutr. 2007 Jan;44(1):63-7. doi: 10.1097/01.mpg.0000239733.79487.1e. PMID 17204955
- [Background] Varni JW, Lane MM, Burwinkle TM, Fontaine EN, Youssef NN, Schwimmer JB, Pardee PE, Pohl JF, Easley DJ. Health-related quality of life in pediatric patients with irritable bowel syndrome: a comparative analysis. J Dev Behav Pediatr. 2006 Dec;27(6):451-8. doi: 10.1097/00004703-200612000-00001. PMID 17164617
- [Background] Christensen MF, Mortensen O. Long-term prognosis in children with recurrent abdominal pain. Arch Dis Child. 1975 Feb;50(2):110-4. doi: 10.1136/adc.50.2.110. PMID 1130815
- [Background] Huertas-Ceballos A, Logan S, Bennett C, Macarthur C. Dietary interventions for recurrent abdominal pain (RAP) and irritable bowel syndrome (IBS) in childhood. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD003019. doi: 10.1002/14651858.CD003019.pub2. PMID 18254014
- [Background] Huertas-Ceballos AA, Logan S, Bennett C, Macarthur C, Martin AE. WITHDRAWN: Pharmacological interventions for recurrent abdominal pain (RAP) and irritable bowel syndrome (IBS) in childhood. Cochrane Database Syst Rev. 2014 Feb 17;2014(2):CD003017. doi: 10.1002/14651858.CD003017.pub3. PMID 24532249
- [Background] American Academy of Pediatrics Subcommittee on Chronic Abdominal Pain; North American Society for Pediatric Gastroenterology Hepatology, and Nutrition. Chronic abdominal pain in children. Pediatrics. 2005 Mar;115(3):e370-81. doi: 10.1542/peds.2004-2523. PMID 15741363
- [Background] Ong DK, Mitchell SB, Barrett JS, Shepherd SJ, Irving PM, Biesiekierski JR, Smith S, Gibson PR, Muir JG. Manipulation of dietary short chain carbohydrates alters the pattern of gas production and genesis of symptoms in irritable bowel syndrome. J Gastroenterol Hepatol. 2010 Aug;25(8):1366-73. doi: 10.1111/j.1440-1746.2010.06370.x. PMID 20659225
- [Background] Carlson MJ, Moore CE, Tsai CM, Shulman RJ, Chumpitazi BP. Child and parent perceived food-induced gastrointestinal symptoms and quality of life in children with functional gastrointestinal disorders. J Acad Nutr Diet. 2014 Mar;114(3):403-413. doi: 10.1016/j.jand.2013.10.013. Epub 2013 Dec 19. PMID 24360501
- [Background] Chumpitazi BP, Cope JL, Hollister EB, Tsai CM, McMeans AR, Luna RA, Versalovic J, Shulman RJ. Randomised clinical trial: gut microbiome biomarkers are associated with clinical response to a low FODMAP diet in children with the irritable bowel syndrome. Aliment Pharmacol Ther. 2015 Aug;42(4):418-27. doi: 10.1111/apt.13286. Epub 2015 Jun 24. PMID 26104013
- [Background] Laird KT, Sherman AL, Smith CA, Walker LS. Validation of the Abdominal Pain Index using a revised scoring method. J Pediatr Psychol. 2015 Jun;40(5):517-25. doi: 10.1093/jpepsy/jsu118. Epub 2015 Jan 22. PMID 25617048
- [Background] Erhart M, Ellert U, Kurth BM, Ravens-Sieberer U. Measuring adolescents' HRQoL via self reports and parent proxy reports: an evaluation of the psychometric properties of both versions of the KINDL-R instrument. Health Qual Life Outcomes. 2009 Aug 26;7:77. doi: 10.1186/1477-7525-7-77. PMID 19709410